CLINICAL TRIAL: NCT00319930
Title: A Phase 1, Multi-Center, Open-Label, Dose-Escalation, Pharmacodynamic Study of Intravenously Administered CNF1010 (17-(Allylamino)-17-demethoxy-geldanamycin [17-AAG]) in Patients With ZAP-70 Positive B-Cell Chronic Lymphocytic Leukemia (CLL)
Brief Title: Phase 1, Dose-Escalation, Pharmacodynamic Study of IV CNF1010 in ZAP-70 Positive CLL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Discontinuation of program
Sponsor: Biogen (Industry)
Responsible Party: Study MD, Biogen Idec
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNF1010-CLL-05001; 110CL101
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2010-03-08 (Estimated); Status verified 2010-03

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic lymphocytic leukemia; CLL; ZAP-70; Hsp90 inhibitor
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — tanespimycin

INTERVENTIONS:
Drug: CNF1010 (17-AAG)

SUMMARY:
The purpose of the study is to evaluate the effects of increasing doses of CNF1010 on pharmacodynamic markers and hematological response.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of B-cell CLL including

   * Lymphocytosis of >=5,000 monoclonal B-cells/microliter co-expressing >= one B-cell marker (CD19, CD20, or CD23) and CD5 in peripheral blood AND
   * <= 55% prolymphocytes AND
   * Bone marrow with >=30% mononuclear cells being lymphocytes
2. ZAP-70 positive CLL
3. Intermediate or High risk, poor prognosis CLL refractory to fludarabine-based therapy as defined by one of the following:

   * Disease progression following 2 cycles of fludarabine OR
   * Failure to achieve PR or CR after at least 2 cycles OR
   * No response to treatment or stable disease after at least 2 cycles of fludarabine OR
   * Disease progression after chemotherapy treatment after fludarabine-based therapy

   OR

   · CLL patients intolerant to fludarabine-based therapy. [Intolerance is defined as the development of any serious medical condition occurring after exposure to fludarabine that would restrict further use of the agent as treatment for the patient's CLL (i.e., autoimmune hemolytic anemia, myelosuppression, hypersensitivity)]
4. Indication for treatment as defined by the NCI Working Group Guidelines
5. Laboratory parameters as follows:

   * Hemoglobin >=10 g/dL (may be post-transfusion); platelet count >=50 x103/mm3
   * T. Bili <2 x ULN and ALT and AST <2 x ULN
   * Creatinine <=2 x ULN
6. ECOG Performance Score <=2
7. For patients of child-producing potential, use of effective contraceptive methods during the study and for 1 month following treatment

Key Exclusion Criteria:

1. Pregnant or nursing women
2. Class III or IV cardiac disease defined by the New York Heart Association Functional Classification and/or left ventricular ejection fraction <40%
3. History of prior radiation that potentially included the heart in the field.
4. History of myocardial infarction or active ischemic heart disease within 6 months of study entry
5. History of arrhythmia (including atrial fibrillation, multifocal premature ventricular contractions, ventricular bigeminy or trigeminy, ventricular tachycardia or a requirement for antiarrhythmics (including digoxin)
6. Baseline QTc >=450 msec for men and >= 470 msec for women in the absence of correctable electrolyte imbalance
7. Poorly controlled angina
8. Congenital long QT syndrome or first-degree relative with unexplained sudden death <40 years of age
9. Presence of left bundle branch block
10. Treatment with chemotherapy, monoclonal antibody or radiotherapy within 28 days of study entry
11. Severe or debilitating pulmonary disease
12. Participation in any investigational drug study within 28 days prior to CNF1010 administration. (Patient must have recovered from all acute effects of previously administered investigational agents)
13. Presence of active malignancy with the exception of basal cell carcinoma
14. Active symptomatic fungal, bacterial and/or viral infection including active HIV or viral (A, B or C) hepatitis
15. Known allergy to soy
16. Requirement for concomitant therapy with drugs that alter metabolism by cytochrome P450 3A4 except low-dose warfarin for implanted device patency
17. Requirement for concomitant therapy with drugs that prolong or may prolong QTc interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-05; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The minimal biologically active dose (MBAD)
Safety and toxicity profile
Pharmacokinetics (PK)
Pharmacodynamics (PD)
Clinical and hematological response

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Ocoee, Florida
  - Albany, New York
  - Dayton, Ohio
  - Greenville, South Carolina
  - Tyler, Texas
  - Norfolk, Virginia